CLINICAL TRIAL: NCT02911610
Title: Open and Controlled Trial to Assess the Arthroscopy Use in Patients Undergoing Wrist Fracture Surgery by Volar Plate
Brief Title: Assessment of Arthroscopy in Patients Undergoing Wrist Fracture
Acronym: WRIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Mª José Perez Úbeda, MD, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16.206_BS
Record Dates: First submitted 2016-06-17; First posted 2016-09-22 (Estimated); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Wrist Injuries
MeSH Terms: conditions — Wrist Injuries | interventions — Arthroscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arthroscopy + volar plate (Experimental): surgery of wrist fractures with volar plate and added arthroscopy
  Interventions: Device: arthroscopy + volar plate
- volar plate (Other): surgery of wrist fractures with volar plate
  Interventions: Device: Volar plate

INTERVENTIONS:
Device: arthroscopy + volar plate — surgery of wrist fractures with volar plate and added arthroscopy
  Arms: Arthroscopy + volar plate
Device: Volar plate — surgery of wrist fractures with volar plate
  Arms: volar plate

SUMMARY:
The use of arthroscopy with the surgery of wrist fractures has a great health and economic impact (prolongs the time of surgery, requires adequately trained personnel, increases the time and surgical expenses and the risk of complications, however, in return ameliorate the prognosis and improves the functional recovery). There are few clinical trials showing a sufficient level of evidence in comparing the results of the surgical treatment of these fractures with volar plate and added arthroscopy so it is necessary to perform a clinical trial with an appropriate design and a sufficient sample size to elucidate the usefulness of arthroscopy in wrist fractures. Therefore, the investigators want to perform an open and controlled clinical trial to adequately analyze the role of arthroscopy in the surgical treatment of wrist fractures in the investigators hospitals.

The main objective of the study is to probe the arthroscopy effectiveness in the functionality of the injured wrist by PRWE (a questionnaire assessing pain and wrist function) between the treatment groups of the trial at 12 months after surgery and for this the investigators plan a phase IV multicenter clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Patients able to read and understand the same consent.
* Patients over 18 years
* Broken wrist surgery with criteria based on the following criteria (must meet all):

  * Patients functionally independent, ie, they can make the purchase without help, categorized according Mackenney or patients who require assisted support by crutches / walker for walking.
  * Radiographic unacceptable reduction after 1 attempted closed reduction in the ER, defined as:

    1. dorsal angulation> 0 °
    2. ulnar variance> 3mm postreduction.
    3. Step articular> 1mm (20)
    4. radial inclination <15 °
  * Patients with unstable fracture.

Exclusion Criteria:

* Type III open fractures of Gustilo and Anderson.
* Bilateral fractures (not acceptable include more than one doll per patient for the analysis of the variables in the study, always choosing the wrist of the dominant hand).
* Fractures associated ipsilateral upper limb affection (except distal ulnar fracture).
* Fracture or serious injury prior ipsilateral wrist.
* Medical criteria that contraindicate surgery.
* Patients with low functional demand, categorized as dependent as Mackenney, ie, they need help to go shopping and do not require assisted support by crutches / walker for walking.
* Patients with tumor lesions secondary processes (eg osteosarcoma, prostate cancer, breast cancer, multiple myeloma), congenital metabolic (eg osteogenesis imperfecta) and others involving themselves poor prognosis associated with disease.
* Women with suspected pregnancy or pregnancy can not participate in this clinical trial because the collection of monitoring data is expected performing radiographic examinations, in case of pregnancy, would be contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Patient-rated Wrist Evaluation (PRWE) questionary score | 12 months after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided